CLINICAL TRIAL: NCT06893393
Title: Bringing Nature Into a Psychiatric Ward: Virtual Travels for Inpatient Care in People With Lived Experience of a Severe Mental Disorder
Brief Title: Virtual Travel Into Nature for Individuals With Lived Experience of Severe Mental Disorders
Acronym: Inpatient VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Super Sublime | Super Splendide (Unknown)
Responsible Party: Principal Investigator, Martin Lepage, Deputy Scientific Director, Douglas Mental Health University Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-927
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Investigate the Use of Virtual Reality in Inpatient Psychiatric Care; Complex Mood Disorders
Keywords: implementation; virtual reality; inpatient psychiatric care; nature; virtual travels; complex mood disorders

STUDY DESIGN:
Intervention Model Description: One group will have access to the virtual reality application Toujours Dimanche alongside their treatment as usual during their hospitalization in psychiatric care, the other will be a control group and will only receive treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toujours Dimanche users (Experimental): Participants who will use the virtual reality application Toujours Dimanche in the context of their hospitalization in psychiatric care. Participants will receive treatment as usual and will be able to use the application at their leisure for a period of 15 days.
  Interventions: Device: Virtual travel-into-nature application Toujours Dimanche
- Control group (No Intervention): Participants will not use the virtual reality application Toujours Dimanche. Will receive treatment as usual.

INTERVENTIONS:
Device: Virtual travel-into-nature application Toujours Dimanche — The use of the virtual travel-into-nature application which features real natural environments from the Eastern Canada area.
  Arms: Toujours Dimanche users

SUMMARY:
The goal of the (observational or clinical) trial is to assess the use of the virtual application Toujours Dimanche for individuals hospitalized in a psychiatric care unit. The main questions it aims to answer are:

* Is it feasible and acceptable for individuals currently hospitalized to use virtual reality during their stay?
* What are the effects on mental health of the virtual reality application in individuals hospitalized in psychiatric care?
* What are the barriers and facilitators of using the virtual reality application in a psychiatric ward from the perspective of service users and health care providers? Researchers will compare virtual reality users to control group (treatment as usual only) to see if the use of the application affects social and emotional well-being in the context of hospitalisation in psychiatry.

In the first phase, participants will:

- Be invited to participate in focus groups to assess their interest in the application.

In the second phase, participants will:

* Complete baseline questionnaires on their connection to nature and social and emotional well-being.
* Use the virtual reality application over a 15 day period alongside treatment as usual.
* Complete post-intervention questionnaires and a survey on their use and opinions of the application.

Healthcare provider feedback phase

- Healthcare providers working on the unit will be invited to share their perception of the impact of implementing the virtual application on the unit through surveys which will be sent by email.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of implementing a virtual reality travel into nature application (Toujours Dimanche) in an inpatient psychiatric unit servicing individuals with complex mood disorders. Via a head mounted device, the application allows individuals to immerse themselves into 360 natural environments and offers the possibility to interact with another individual through a private platform. Recruitment will take place on a psychiatric inpatient unit dedicated to individuals with complex mood disorders (e.g. bipolar disorder, unipolar depression). Flyers will be posted at the unit to recruit people hospitalized. Participants with lived experience will also be recruited through the reference of their health care providers at the unit (i.e. treating psychiatrists or other members of the staff). In all cases, the health care provider will obtain the clients' consent prior to being contacted by the research assistant. The research assistant will then meet the prospective participant in person at the unit to explain the research project (inclusion criteria, the consent and assessment procedures, and the application if the participant is interested in being included in the active group) and answer any questions or concerns. Each participant will be presented with the consent form. Additionally , we plan on organizing short presentations to the people hospitalized at the unit. Given the short-term hospitalization at the unit, the researchers want people to hear about the project, but also being able to ask their questions directly to the research team.

For health care providers, they will be recruited through staff meetings. The research coordinator will present the project to professionals during staff meetings and flyers will be posted at the nursing station.

Data Collection and Analysis:

The connectedness to nature scale (CNS) (Mayer & Frantz, 2004) will be administered at baseline only. The CNS is a 14 self-report item questionnaire that assesses individuals' trait levels of feeling emotionally connected to the natural world. The researchers expect that each participant will have a different perspective toward nature that could influence the potential use and effect of the application. The following questionnaires will be administered both at baseline and post-test. The Beck Anxiety Scale (BAI; (Beck et al., 1988)) is a self-report questionnaire that includes 21 items rated on a Likert scale of 0 (not at all) to 3 (Severely). Given that the goal of the Toujours Dimanche application is to reduce stress, the researchers believe it is important to measure anxiety before and after using the application. The BAI has adequate psychometric properties and is a well-recognized scale that encompasses the cognitive, emotional, and physical components of anxiety. The Kessler Psychological Distress Scale (K10) (Kessler et al., 2002) is a 10-item self-report questionnaire assessing distress through questions about anxiety and depression. The 10 items are rated on a Likert scale ranging from 1 (None of the time) to 5 (All the time). Regarding stress, the researchers included the Perceived Stress Scale (PSS), a 10-item self-report questionnaire assessing subjective stress using a Likert scale from 1 (never) to 5 (very often) (Cohen & Williamson, 1988). For the current study, the questionnaire will be modified to adjust the timeframe for the assessment of perceived stress from one month to two weeks. For depressive symptoms, the PHQ-9 (Kroenke et al., 2001) will be used. This 9-item self-report questionnaire assesses depressive symptoms in the last two weeks, rated on a Likert scale ranging from 0 (not at all) to 3 (nearly every day) and has good psychometric properties (Kroenke et al., 2001). Wellbeing will be assessed with the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) (Tennant et al.2007), a 14-item self-report questionnaire using a Likert scale from 1 (never) to 5 (all the time) with good psychometric properties (Lloyd et al., 2012). This scale assesses wellbeing with an holistic approach in the last two weeks. Social isolation will be assessed through a measure of loneliness, and more specifically with the De Jong Gierveld Loneliness Scale - short version (DJGLS) (Gierveld & Tilburg, 2006). This 6-item self-report questionnaire assess overall, emotional, and social loneliness using a Likert scale ranging from 0 (not lonely) to 11 (extremely lonely).

At post-test, the research team will conduct a short semi-structured interview regarding the active group participants' opinion on the application as well as the barriers and facilitators to use it. The audio of this interview will be recorded (as specified in the consent form). The interview will then be transcribed and deleted. Psychiatric diagnosis, medication, duration of illness as well as the number and duration of hospitalizations will be collected from participants' medical records. The participants' consent to access personal information will be asked beforehand (non-mandatory), as part of the informed consent procedure. All measures of baseline will be administered in person at the unit. At post-test, the assessment will be conducted in person at the unit if the participant is still hospitalized. If the person was discharged from the unit, the participant will have the choice to complete the assessment in person at the Douglas, or remotely.

In addition to the outcomes selected by the participant, the researchers will also assess the following objective indicators regarding their use of the application:

* Number of VR sessions completed
* Duration of VR sessions
* Reasons to stop using the application (e.g. not interested, hospital stay is over, etc.)
* Difficulties reported using the application or the VR headset
* Frequency of connection with a relative or the peer helper in the application
* Safety of the study (including whether there are any adverse events reported)

The health care providers will be assessed via an online survey that will last approximately 30 minutes. To access the survey, the health care providers will use the QR code provided on the flyer at the nursing station. Before starting the survey, they will be asked to confirm that they are offering direct care to people hospitalized at the unit (inclusion criterion). Once confirmed, the consent form will be presented, and the health care providers will have to consent electronically. Once this is done, the participants will complete a short sociodemographic questionnaire as well as questions regarding their opinion on the use of the application Toujours Dimanche at the unit, including the barriers and facilitators that they observed for its implementation. For all data from the questionnaires and outcome measures of people with lived experience, they will be entered into Redcap and analyzed using SPSS (IBM SPSS Statistics for Windows. Armonk, NY: IBM Corp). We are also committed to upholding EDI principles rigorously throughout all project phases, including recruitment. SuperSublime is designed to be an inclusive project, welcoming individuals from diverse backgrounds to participate. Several measures are in place to enhance data quality and reduce the likelihood of missing data occurrence. Once data entry into Redcap has been completed, it will be reviewed for quality (e.g., human error) by a second member of the research team. For the online survey completed by the health care providers, the participants will receive a direct Redcap link to complete the questionnaires. All quantitative data files will be stored on the Douglas institutional server. These files will have codes for identification (pseudonyms) and will be password protected.

A list connecting participant names to their pseudonyms will be kept separate from the rest of the data, in a locked filing cabinet in the researcher's office, and in a separate, password-protected electronic file on the institutional server that will only be accessible by the primary researcher and research assistant working on this project.

While using the application, the participant with lived experience and their relatives will access semi-private virtual spaces accessible only by individuals and not by the institution to promote confidentiality. Further, the participants will use their participant ID to access the virtual spaces.

The researchers will use descriptive statistics to summarize sociodemographic and clinical characteristics of the sample. Dependent t-tests will be used to compare the characteristics and scores between the active and the control groups at baseline. Wilcoxon signed-rank tests will be used if the normality assumption is not met for the distribution of the different variables. The total score from the CNS, the answers regarding previous use of VR (sociodemographic questionnaire), the presence of cybersickness symptoms as well as significant differences in baseline variables at baseline will be used as covariates in our analyses to assess their influence on the effect of Toujours Dimanche on the different outcomes, as well as on the use of the application by the participants. Linear mixed models for repeated measures will be used to assess the effect of Toujours Dimanche between groups on the different outcomes with fixed effects of time. Further, answers from the short semi-structured interview will be entered in QDA Miner to assess emergent themes about the application at post-test. Descriptive statistics will be used to summarize the different variables linked to the use of the application (e.g. duration of session, number of sessions).

Further, the barriers and facilitators associated with the use of Toujours Dimanche and VR at the unit will be summarized using descriptive statistics and thematic analyses for both people with lived experience and health care providers.

The researchers aim at recruiting 80 participants with lived experience (40 in the active group and 40 in the control group) to obtain sufficient statistical power using linear mixed models for repeated measures to assess the effect of Toujours Dimanche on the different outcomes with fixed effects of time (power = 0.80, significance level = 0.05, small to medium effect size). Further, to assess the barriers and facilitators from the health care providers' perspective, the researchers aim at recruiting 10 participants to obtain the opinion of different individuals as well as different professions that might have experienced the use of Toujours Dimanche differently.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older
* Being hospitalized in a psychiatric unit at the time of the study
* Being relatively clinically stable, according to the treating psychiatrist
* Being free of uncorrected visual impairments
* Being able to speak or read French or English

Exclusion Criteria:

* Current photosensitive epilepsy or a history of seizures
* Previous history of severe motion sickness or cyber-sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Change from baseline (15 days post)
  The Perceived Stress Scale (PSS), a 10-item self-report questionnaire assessing subjective stress using a Likert scale from 1 (never) to 5 (very often) (Cohen & Williamson, 1988). For the current study, the questionnaire will be modified to adjust the timeframe for the assessment of perceived stress from one moth to two weeks.
Kessler Psychological Distress Scale | Change from baseline (15 days post)
  The Kessler Psychological Distress Scale (K10) (Kessler et al., 2002) is a 10-item self-report questionnaire assessing distress through questions about anxiety and depression. The 10 items are rated on a Likert scale ranging from 1 (None of the time) to 5 (All the time).
Beck Anxiety Scale | Change from baseline (15 days post)
  The Beck Anxiety Scale (BAI; (Beck et al., 1988)) is a self-report questionnaire that includes 21 items rated on a Likert scale of 0 (not at all) to 3 (Severely).
The connectedness to nature scale | Change from baseline (15 days post)
  The connectedness to nature scale (CNS) (Mayer & Frantz, 2004) is a 14 self-report item questionnaire that assesses individuals' trait levels of feeling emotionally connected to the natural world.
PHQ-9 | Change from baseline (15 days post)
  Depressive symptoms will be assessed using the PHQ-9. This 9-item self-report questionnaire assesses depressive symptoms in the last two weeks, rated on a Likert scale ranging from 0 (not at all) to 3 (nearly every day)
Warwick-Edinburgh Mental Well-being Scale | Change from baseline (15 days post)
  Wellbeing will be assessed with the Warwick-Edinburgh Mental Well-being Scale (WEMWBS), a 14-item self-report questionnaire using a Likert scale from 1 (never) to 5 (all the time).
De Jong Gierveld Loneliness Scale - short version | Change from baseline (15 days post)
  Social isolation will be assessed with the De Jong Gierveld Loneliness Scale - short version (DJGLS). This 6-item self-report questionnaire assess overall, emotional, and social loneliness using a Likert scale ranging from 0 (not lonely) to 11 (extremely lonely).

CONTACTS AND LOCATIONS:
Overall Officials: Élisabeth Thibaudeau, Ph.D., Principal Investigator — Laval University
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The data from this project are collected with people hospitalized in only one specific unit at the Douglas hospital and sharing their individual data might comprise their confidentiality.

REFERENCES:
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Gierveld JDJ, Tilburg TV. A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Research on Aging 2006;28(5):582-598.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- See also: Company website for the company responsible for the creation of the virtual travel-into-nature application Toujours Dimanche — https://www.supersplendide.com/